CLINICAL TRIAL: NCT06307249
Title: Precision Therapy for Solid Tumors: Synergistic Inhibition of Cell Proliferation and Angiogenesis Via CDK4/6 and Anti-VEGF Approach Targeting LncRNA Expression
Brief Title: Precision Therapy for Solid Tumors: Synergistic CDK4/6 Inhibition and Anti-VEGF Targeting LncRNA
Acronym: PTST_PALBEVA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lebanese University (Other)
Collaborators: Haykel Hospital (Unknown)
Responsible Party: Principal Investigator, Nehman Makdissy, Principal Investigator, Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LU_HH_Cancer_Precision Therapy
Record Dates: First submitted 2024-02-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Solid Tumor; Colorectal Cancer; Breast Cancer; Ovarian Cancer; Lung Cancer; Targeted Therapy; Chemotherapy; Immunotherapy; Precision Therapy
Keywords: LncRNA; Anti-VEGF; CDK4/6 inhibitor; Gene Polymorphism; Palbociclib; Bevacizumab; Inflammation; Immune Cells; Angiogenesis; Proliferative; Cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Inflammation | interventions — palbociclib; Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Carrier First-line Combined Therapy Group C-FL-CT (Experimental): This group of patients, who are carriers of the risk alleles, will receive combined therapy as the initial first-line treatment without prior chemotherapy.
  Interventions: Genetic: SNP; Drug: Palbociclib 125mg; Drug: Bevacizumab
- Carrier Second-line Combined Therapy Group C-SL-CT (Experimental): This group of patients, who are carriers of the risk alleles, will receive combined therapy after having undergone prior chemotherapy, making it the second-line treatment.
  Interventions: Genetic: SNP; Drug: Palbociclib 125mg; Drug: Bevacizumab
- Non-carrier First-line Combined Therapy Group NC-FL-CT (Experimental): This group of patients, who are non-carriers of the risk alleles, will receive combined therapy as the initial first-line treatment without prior chemotherapy.
  Interventions: Genetic: SNP; Drug: Palbociclib 125mg; Drug: Bevacizumab
- Non-carrier Second-line Combined Therapy Group NC-SL-CT (Experimental): This group of patients, who are non-carriers of the risk alleles, will receive combined therapy after having undergone prior chemotherapy, making it the second-line treatment.
  Interventions: Genetic: SNP; Drug: Palbociclib 125mg; Drug: Bevacizumab

INTERVENTIONS:
Genetic: SNP — Diagnostics of patients' carriers or not of the risk allele(s)
  Other Names: Risk Allele(s)
Drug: Palbociclib 125mg — Palbociclib 125mg/day/os over 21 days every 28 days
  Other Names: anti-CDK4/6
Drug: Bevacizumab — 10mg/kg every 21 days
  Other Names: Anti-VEGF

SUMMARY:
Solid tumors pose significant challenges in current therapeutic approaches. Targeted therapy has emerged as a promising avenue, aiming to enhance treatment efficacy while minimizing adverse effects. This clinical trial focuses on an innovative combination of two targeted inhibitors, Palbociclib and Bevacizumab, for their potential synergistic effects in addressing these challenging malignancies. Moreover, this study incorporates a molecular approach by considering Long Non-Coding RNAs (LncRNAs) as biomarkers. Initiating with a focus on colorectal cancer, the study aims to expand its scope to other solid tumors, including lung, breast, ovarian and other cancers. Palbociclib, a cyclin-dependent kinase 4/6 (CDK4/6) inhibitor, disrupts the cell cycle progression, particularly in cancer cells with specific molecular characteristics. Bevacizumab, a vascular endothelial growth factor (VEGF) inhibitor, targets angiogenesis-a critical process for tumor growth and metastasis. The rationale behind combining these agents lies in their complementary mechanisms of action, potentially leading to enhanced antitumor effects. LncRNAs have shown promise in predicting treatment response and prognosis in various cancers, providing an additional layer of precision to the treatment strategy. By elucidating the molecular basis through LncRNA analysis, the trial aims to tailor the treatment to the specific molecular profile of each patient, ultimately striving for better outcomes and improved survival rates. This novel combination therapy, coupled with a personalized biomarker-driven approach, represents a cutting-edge strategy in the pursuit of more effective and individualized treatment for solid tumors.

DETAILED DESCRIPTION:
This innovative clinical trial applies a comprehensive strategy to study the complex interplay of biomarkers, immune responses, angiogenesis, and proliferation in solid tumor progression. This approach integrates the selective cyclin-dependent kinase 4/6 (CDK4/6) inhibitor, such as Palbociclib, with the angiogenesis inhibitor, like Bevacizumab. This dual-targeted therapy holds promise for treating various solid tumors, including colorectal cancer, breast cancer, lung cancer, ovarian cancer, and others.

A focal point of the study is the investigation of Long Non-Coding RNA (LncRNA) , chosen for its potential as a prognostic and predictive biomarker. LncRNA plays a multifaceted role in cellular processes, influencing cell cycle checkpoints, angiogenesis, and metastasis. Its aberrant expression across different cancers positions as a key subject of investigation, particularly considering its potential association with polymorphisms. Beyond its involvement in proliferation and angiogenesis. It also adds an additional layer of complexity, crucial for understanding patient outcomes.

The investigation initiates with colorectal cancer and extends to other solid cancers, including lung, ovarian, and breast cancers. Patients are stratified into carriers or non-carriers of the risk allele, forming the foundation for precision-driven treatments. The study design comprises two distinct groups within the colorectal cancer cohort, Group 1 and Group 2, involving patients with and without the risk allele. These groups undergo combined therapy with a CDK4/6 inhibitor and anti-VEGF. Similarly, the distribution is maintained for patients with and without the risk allele in other solid tumors (lung, breast, ovarian, etc.), receiving the same combined therapy tailored to their molecular profiles whether taken as 1st line of treatment or 2nd line of treatment.

Precise pre-treatment assessments establish baseline parameters, while post-treatment evaluations cover outcomes such as tumor progression, cancer regression, survival rates, and thromboembolic events. The interdependent relationship between proliferative tumor cells and angiogenesis, coupled with the potential impact of thromboembolism, is pivotal for cancer progression. Dysregulated cell cycle machinery, often involving overactive cyclin-dependent kinases (CDKs) like CDK4/6, drives uncontrolled proliferation, leading to a hypoxic microenvironment that triggers angiogenesis. Recognizing this symbiosis, the rationale for combining Palbociclib, a CDK4/6 inhibitor, with Bevacizumab, an anti-VEGF agent, becomes evident. While Palbociclib disrupts the cell cycle progression of proliferating tumor cells, hindering their uncontrolled growth, Bevacizumab concurrently targets the angiogenic process by inhibiting VEGF.

This dual-targeted approach aims to comprehensively address both the proliferative, angiogenic, and thromboembolic facets of tumor biology, potentially leading to a more effective and synergistic anti-tumor response.

Four groups will be considered:

Carrier Groups:

Group 1: "Carrier First-line Combined Therapy Group", C-FL-CT; Group 2: "Carrier Second-line Combined Therapy Group", C-SL-CT

Non-carrier Groups:

Group 3: "Non-carrier First-line Combined Therapy Group", NC-FL-CT; Group 4: "Non-carrier Second-line Combined Therapy Group", NC-SL-CT "Carrier"" denotes the patient who possesses the risk allele of the LncRNA CDKN2B-AS1.

Group 1: This group of patients, who are carriers of the risk alleles, will receive combined therapy as the initial first-line treatment without prior chemotherapy.

Group 2: This group of patients, who are carriers of the risk alleles, will receive combined therapy after having undergone prior chemotherapy, making it the second-line treatment.

Group 3: This group of patients, who are non-carriers of the risk alleles, will receive combined therapy as the initial first-line treatment without prior chemotherapy.

Group 4: This group of patients, who are non-carriers of the risk alleles, will receive combined therapy after having undergone prior chemotherapy, making it the second-line treatment.

In summary, the study integrates precision medicine, biomarker-driven therapies, and a comprehensive understanding of the molecular basis of tumor progression, including thromboembolism. This approach offers a promising avenue for the development of personalized and effective treatments for various solid tumors, emphasizing not only efficacy and safety but also the overall effectiveness of the proposed therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of white ethnicity.
* Age between > 18
* Both males and females.
* Diagnosis of selected cancer type (e.g., colorectal cancer, lung cancer, genitourinary cancers, breast cancer).
* Cancer stage III/ IV with or without metastasis or lymph node dissemination at the time of enrollment.
* Unrelated patients.

Exclusion Criteria:

* History of hematological cancer types or previous cancers, recurrent or relapse.
* Diagnosis of inflammatory bowel diseases.
* Pre-existing cardiovascular diseases or coronary artery diseases.
* Confirmed treated or untreated autoimmune diseases.
* Metabolic disorders, diabetes, or hypertension.
* Neurological diseases.
* Evidence of cardiac, renal, bone, or cerebral damage.
* Presence of more than one type of malignancies.
* Active infections or myositis.
* Familial polyposis.
* Alcohol or smoking habits.
* Body mass index (BMI) >30.
* Significant weight loss within the last 2 years.
* History of surgeries.
* Pregnancy.
* Related patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Cancer Progression | [Time Frame: up to 60 months]
  The assessment of cancer progression will be conducted using the standardized TNM staging system and applying the Response Evaluation Criteria (RECIST) guideline (ver. 1.1). Progression-Free Survival (PFS), a key primary clinical endpoint for assessing cancer progression, will be calculated as the duration (in months) from the date of enrollment in the study until the tumor progresses, new lesions appear, or until the participant's death from any cause based on RECIST guidelines, considering an increase in tumor size or the appearance of new lesions according to imaging assessments (e.g., CT, MRI, or PET scans) and clinical evaluations (including tumor markers and histopathological analysis).
Identification of Potential Biomarkers | [ Time Frame: Once at the moment of the patient's enrollment in the study]
  Finding and characterizing new biomarkers linked to thromboembolism and the advancement of cancer is the aim of this result. The evaluation will pay particular attention to Long Non-Coding RNAs (LncRNAs). At the time of study enrollment, biological samples (such as blood or tissue) from enrolled patients will be collected as part of the identification procedure. With Ct (Cycle threshold) serving as the standard unit of measurement for all genes, the evaluation will employ quantitative PCR (qPCR) to study and assess the expression and polymorphisms of the investigated genes. This thorough evaluation seeks to further our knowledge of the molecular markers and the course of cancer, shedding light on new pathways for diagnosis and treatment that might lead to better patient outcomes
Evaluation of Treatment Response to Palbociclib and Bevacizumab Combination Therapy | [ Time Frame: up to 60 months]
  This main outcome evaluates the extent to which patients responding to combination therapy are managing both angiogenesis and the cancer cell cycle progression. The percentage change in tumor size, a measure of therapy efficacy, will be calculated using the RECIST criteria in the evaluation.

SECONDARY OUTCOMES:
Survival Rates | [ Time Frame: up to 60 months]
  Analysis of overall survival and progression-free survival rates among groups
Adverse Events | [ Time Frame: up to 60 months]
  Monitoring and reporting of adverse events related to the Palbociclib and Bevacizumab treatment regimen.
Assessment of Immune Checkpoint Expression (e.g., PD-1 and CTLA-4) | [ Time Frame: up to 60 months]
  The expression of immunological checkpoint molecules, namely cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) and programmed cell death protein 1 (PD-1) is the main emphasis of this result. The goal is to comprehend how immunological checkpoints control the immune response. PCR or flow cytometry will be used to determine immunological checkpoint expression as part of the evaluation. The percentage of change in PD-1 and CTLA-4 expression levels throughout a 60-month period in comparison to their levels at the diagnostic time will be used to measure the results. Over the course of the study, a thorough knowledge of the immune checkpoint dynamics and their influence on the immune response is made possible by the consistent evaluation that is ensured by the use of a standardized common unit of measure.
Measurement of Angiogenic Factors (e.g., VEGF) | [ Time Frame: up to 60 months]
  This study aims to evaluate the angiogenic factor Vascular Endothelial Growth Factor (VEGF) post-treatment. VEGF plays a crucial role in regulating angiogenesis and is linked to tumor vascularization. The serum concentrations of VEGF-A/C will be measured by ELISA, providing valuable insights into the angiogenic processes linked to the treatment outcomes.
Measurement of Tumor Proliferation Markers (e.g., Ki67, P16) | [ Time Frame: up to 60 months].
  The study incorporates the evaluation of tumor proliferation markers, including Ki67 a protein present in active phases of cell cycle and P16 a tumor suppressor protein, utilizing assays of immunohistochemistry (IHC) to measure the expression levels of Ki67 and P16 (in percent %). These assays play a pivotal role in quantifying the extent of tumor cell division, giving valuable insights into the rate of tumor growth. This comprehensive analysis of proliferation markers aims to enhance our understanding of the tumor's behavior upon the therapeutic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, Professor, Study Chair — Lebanese University
Locations (2):
- Lebanon (2):
  - Haykel Hospital, Tripoli, North Lebanon
  - Lebanese University, Tripoli, North Lebanon

IPD SHARING:
Plan to Share IPD: No